CLINICAL TRIAL: NCT03516500
Title: This is a Phase II Study on the Safety and Feasibility of Identifying the Intersegmental Plane of the Lung by Iron Sucrose Injection Staining,Both on the Pleural Surface and Lung Parenchyma
Brief Title: Trial of Identifying the Lung Intersegmental Plane by Iron Sucrose Injection Staining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Head of Thoracic Surgery, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-006
Record Dates: First submitted 2018-03-30; First posted 2018-05-04 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Lung Neoplasm; Segmentectomy;Intersegmental Plane
MeSH Terms: conditions — Lung Neoplasms | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Intervention Model Description: After the investigators cut the pulmonary vessels and ligate the segmental bronchus. The investigators inject Iron Sucrose (100 mg dissolved in 50 mL saline) through a butterfly needle into the bronchus of the targeting segment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iron Sucrose injection group (Experimental): The investigators inject Iron Sucrose (100 mg dissolved in 50 mL saline) through a butterfly needle into the bronchus of the targeting segment.
  Interventions: Drug: Iron Sucrose Injection

INTERVENTIONS:
Drug: Iron Sucrose Injection — The investigators inject Iron Sucrose (100 mg dissolved in 50 mL saline) into the segmental bronchus.

SUMMARY:
This is a protocol to determine the safety and feasibility of using Iron Sucrose Injection to identify the intersegmental plane,not only on the pleural surface but also the parenchyma of the lung.

DETAILED DESCRIPTION:
This is a protocol to determine the safety and feasibility of using Iron Sucrose Injection to identify the lung intersegmental plane. This is relevant because the detection of small and early lung cancer is becoming increasingly common. segmentectomy may become a more prominent procedure for early-small lung cancer. One of the most difficult aspects of complete segmentectomy is detection of the intersegmental plane while maintaining an adequate surgical margin and remaining lung function. The method used to detect the intersegmental plane remains controversial. It is hoped that this technology can be used to recognize the intersegmental plane on the pleural surface and the pulmonary parenchyma and will save lots of money for patients in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤age ≤80 years
* The patient must be scheduled to undergo segmentectomy or combined subsegmentectomy.
* The patient must be willing and able to comply with all study requirements and have understood and signed the informed consent.

Exclusion Criteria:

* A known allergy to Iron Sucrose Injection
* The patients who have Iron overdose or iron utilization barrier Intra-operative founding of extensive pigmentation Silicosis or extensive carbon deposition in the lung.
* Patients who have not received segmental resection.
* Patients who converted to thoracotomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related grade 3-5 adverse events | Up to 90 days post-surgery
  Incidence of treatment-related grade 3-5 adverse events assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0

SECONDARY OUTCOMES:
Surgical margin | Day of surgery
  Intraoperative measured by the surgeons.From the tumor peripheral to the lung margin.According to the guidelines,the margins should ≥2cm or ≥ the size of the tumor.

OTHER OUTCOMES:
duration of air leaks | 30 days after the patient was discharged.
  when there is no air leak in the drainage system
Hospital Costs | 30 days after the patient was discharged
  The expenses incurred in hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The investigators hope the data will available in the end of 2018.

REFERENCES:
- [Derived] Li C, Zhang X, Feng X, Han D, Xiang J, Li H. A feasible technique for distinguishing the intersegmental plane by transbronchial injection of iron sucrose. JTCVS Tech. 2023 Jan 16;18:137-142. doi: 10.1016/j.xjtc.2022.12.007. eCollection 2023 Apr. PMID 37096093